CLINICAL TRIAL: NCT02613234
Title: Efficacy of 128-channel Electroencephalograph Combined With BESA Dipole Localization Method and Intervention on Brain Waves for Epilepsy
Brief Title: Efficacy of 128-channel EEG Combined With BESA Dipole Localization and Intervention on Brain Waves for Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Weifeng Peng, Vice Professor, Neurology Department, Investigator, Clinical Doctor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 128EEG
Record Dates: First submitted 2015-11-15; First posted 2015-11-24 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; 128-Channel EEG; Dipole Localization; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Active Intervention on brain waves by cathode tDCS
  Interventions: Device: cathode tDCS
- Control Group (Sham Comparator): Sham Intervention on brain waves by cathode tDCS
  Interventions: Device: Sham cathode tDCS

INTERVENTIONS:
Device: cathode tDCS — At the first randomized controlled stage, the experimental group will undergo five daily sessions of active brain-wave intervention by cathode tDCS (20min, 1mA) targeting the epileptogenic focus, which is confirmed by 128-channel EEG and BESA dipole localization method.
  At the second open-label extension stage, all the patients will undergo five daily sessions of active intervention (20min, 1mA).
  Arms: Experimental Group
Device: Sham cathode tDCS — At the first randomized controlled stage, the control group will undergo five daily sessions of sham brain-wave intervention by cathode tDCS (20min, 1mA, the stimulator will be turned off after 5s) targeting the epileptogenic focus, which is confirmed by 128-channel EEG and BESA dipole localization method.
  At the second open-label extension stage, all the patients will undergo five daily sessions of active intervention (20min, 1mA).
  Arms: Control Group

SUMMARY:
The prevalence of epilepsy is about 0.5% to 1% worldwide, with high disability and mortality rate. The 128-channel electroencephalograph (EEG), combined with BESA dipole localization method, is able to provide more specific information about the brain activity and find out the epileptogenic focus. Based on this novel EEG recording method, cathode transcranial direct current stimulation (tDCS) targeting the epileptogenic focus can be used to decrease the excitability of the cortex, thus reducing the frequency of seizures. A single-center double-blinded randomized controlled and open-label extension trial will be carried out to study the efficacy of 128-channel electroencephalograph combined with BESA dipole localization method and Intervention on brain waves for epilepsy.

DETAILED DESCRIPTION:
Background: The prevalence of epilepsy is about 0.5% to 1% worldwide, with high disability and mortality rate. The 128-channel electroencephalograph (EEG), combined with Brain Electrical Source Analysis (BESA) dipole localization method, is able to provide more specific information about the brain activity and find out the epileptogenic focus. Based on this novel EEG recording method, cathode transcranial direct current stimulation (tDCS) targeting the epileptogenic focus can be used to decrease the excitability of the cortex, thus reducing the frequency of seizures.

Methods: A single-center double-blinded randomized controlled and open-label extension trial will be carried out to study the efficacy of 128-channel electroencephalograph combined with BESA dipole localization method and Intervention on brain waves for epilepsy. Adult patients aged 18 to 65 years old with epilepsy will be recruited. The study contains two stages. At the first randomized controlled stage, patients will be randomly assigned to experimental and control group with a 1:1 sqrt allocation and undergo five daily sessions of brain-wave intervention by cathode tDCS （20min, 1mA） targeting the epileptogenic focus, which is confirmed by 128-channel EEG and BESA dipole localization method. Active intervention will be carried out for the experimental group, and sham intervention ( the stimulator will be turned off after 5s) for the control group. The frequency of seizures, the number of epileptiform discharges, the diffusion tensor imaging (DTI) of magnetic resonance imaging (MRI), the cognitive function, the psychology and the life quality will be measured before (baseline), 1 hour, 4 weeks and 12 weeks after the last intervention to evaluate the changes after intervention. At the second open-label extension stage, all the patients will undergo five daily sessions of active intervention (20min, 1mA) and be followed up for 12 weeks similar to the first stage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with epilepsy at least 1 year according to the 2010 International League Against Epilepsy (ILAE) criteria.
* Aged 18 to 65 years old.
* The seizure is not well-controlled by antiepileptic drugs, the patient cannot tolerant the side effect of antiepileptic drugs, or the patient is not satisfied with the curative effect.
* The dose of antiepileptic drugs must be stable in the last 4 weeks.
* The patient or his/her family member is able to recording the frequency of seizures and complete the trial.

Exclusion Criteria:

* History of status epilepticus in the last 12 weeks according to the definition by Neurocritical Care Society (NCS) 2012.
* History of transcranial direct current stimulation, repetitive transcranial magnetic stimulation, vagus nerve stimulation, trigeminal nerve stimulation or deep brain stimulation. History of pacemaker or other metal equipment implantation.
* History of skull defect, brain tumor, encephalitis, progressive encephalopathy and other progressive diseases of central nervous system.
* History of severe cardiac, hepatic, renal, hematologic diseases, or other progressive and systemic diseases, or during pregnancy.
* History of major depression and other mental disturbance, color blindness, hearing or language disorder who is not able to complete the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | 6 months
  The frequency of seizures using diary

SECONDARY OUTCOMES:
MMSE | 6 months
  The cognitive function using Mini-mental state examination
MoCA | 6 months
  The cognitive function using Montreal cognitive assessment
AVLT | 6 months
  The cognitive function using auditory verbal learning test (
SDMT | 6 months
  The cognitive function using symbol digit modalities test
CWT | 6 months
  The cognitive function using Stroop color word test
EPQ | 6 months
  The psychology evaluation using Eysenck personality questionnaire
HAMD-17 | 6 months
  The psychology evaluation using Hamilton rating scale for depression-17
SCL-90 | 6 months
  The psychology evaluation using symptom check list-90
QOLIE-31 | 6 months
  The life quality using quality of life in epilepsy-31
Epileptiform discharges | 6 months
  The number of epileptiform discharges using 30min EEG
fMRI analysis | 6 months
  Graph theory-based fMRI analysis

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Department of Neurology, Zhongshan Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China